CLINICAL TRIAL: NCT07228819
Title: Sustainability Via Active Garden Education (SAGE): Scaling up Evidence-based, Policy-guided Physical Activity and Nutrition Education for Preschoolers
Brief Title: Sustainability Via Active Garden Education Wellness Implementation Strategies in Early Care and Education
Acronym: SAGE WISE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Penn State University (Other); Texas A&M University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rebecca Lee, Professor, Arizona State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022025; R01HD116828-01 (NIH)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Implementation Science; Diet, Food, and Nutrition; Child Care; Motor Behavior
Keywords: Child; Preschool; Nutrition; Exercise; Health; Policy; School; Garden
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental: (S1) E-support, (S2) in-person support, (S3) Learning collaborative (Experimental): Schools will receive all three strategies: (S1) e-support implementation package which comprises the SAGE basic with the additional e-support implementation package that includs semi-weekly teacher text messages, a weekly check in phone call, and a teacher hotline. (S2) in person staff support and teacher training which requires SAGE curriculum activities to be completed in a single session to accommodate research staff schedules. (S3) virtual learning collaborative which will be developed in consultation with an advisory board with the goal of increasing the social network connectivity and community capacity about garden-based outdoor learning in preschoolers. ECE sites assigned to this condition will receive access to the original SAGE basic plus an online portal (such as a moderated Facebook private group) where they will be able to share information and interactions about garden learning. Monthly implementation "tips and tricks" video
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE e-support; Behavioral: SAGE in-person support; Behavioral: Learning collaborative
- (S1) E-support, (S2) in-person support (Experimental): Schools will receive all two of the three strategies: (S1) e-support implementation package which comprises the SAGE basic with the additional e-support implementation package that includs semi-weekly teacher text messages, a weekly check in phone call, and a teacher hotline. (S2) in person staff support and teacher training which requires SAGE curriculum activities to be completed in a single session to accommodate research staff schedules.
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE e-support; Behavioral: SAGE in-person support
- (S3) Learning collaborative, (S2) in-person support (Experimental): Schools will receive two strategies: (S2) in person staff support and teacher training which requires SAGE curriculum activities to be completed in a single session to accommodate research staff schedules. (S3) virtual learning collaborative which will be developed in consultation with an advisory board with the goal of increasing the social network connectivity and community capacity about garden-based outdoor learning in preschoolers. ECE sites assigned to this condition will receive access to the original SAGE basic plus an online portal (such as a moderated Facebook private group) where they will be able to share information and interactions about garden learning. Monthly implementation "tips and tricks" video
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE in-person support; Behavioral: Learning collaborative
- (S2) in-person support (Experimental): Schools will receive all one strategy: (S2) in person staff support and teacher training which requires SAGE curriculum activities to be completed in a single session to accommodate research staff schedules.
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE in-person support
- Control (Experimental): Schools will receive SAGE baseline curriculum access and study materials.
  Interventions: Behavioral: SAGE Basic
- (S1) E-support, (S3) Learning collaborative (Experimental): Schools will receive all two strategies: (S1) e-support implementation package which comprises the SAGE basic with the additional e-support implementation package that includs semi-weekly teacher text messages, a weekly check in phone call, and a teacher hotline. (S3) virtual learning collaborative which will be developed in consultation with an advisory board with the goal of increasing the social network connectivity and community capacity about garden-based outdoor learning in preschoolers. ECE sites assigned to this condition will receive access to the original SAGE basic plus an online portal (such as a moderated Facebook private group) where they will be able to share information and interactions about garden learning. Monthly implementation "tips and tricks" video
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE e-support; Behavioral: Learning collaborative
- (S1) E-support (Experimental): Schools will receive all one strategy: (S1) e-support implementation package which comprises the SAGE basic with the additional e-support implementation package that includes semi-weekly teacher text messages, a weekly check in phone call, and a teacher hotline.
  Interventions: Behavioral: SAGE Basic; Behavioral: SAGE e-support
- (S3) Learning collaborative (Experimental): Schools will receive one strategy: (S3) virtual learning collaborative which will be developed in consultation with an advisory board with the goal of increasing the social network connectivity and community capacity about garden-based outdoor learning in preschoolers. ECE sites assigned to this condition will receive access to the original SAGE basic plus an online portal (such as a moderated Facebook private group) where they will be able to share information and interactions about garden learning. Monthly implementation "tips and tricks" video
  Interventions: Behavioral: SAGE Basic; Behavioral: Learning collaborative

INTERVENTIONS:
Behavioral: SAGE Basic — SAGE basic includes installation/refresh of an ECE garden, 12 lesson curriculum with delivery materials.
Behavioral: SAGE e-support — Semi-weekly teacher text messages, a monthly newsletter and a teacher hotline
  Arms: (S1) E-support; (S1) E-support, (S2) in-person support; (S1) E-support, (S3) Learning collaborative; Experimental: (S1) E-support, (S2) in-person support, (S3) Learning collaborative
Behavioral: SAGE in-person support — Weekly in person support and training following the "see one, do one, teach one" model
  Arms: (S1) E-support, (S2) in-person support; (S2) in-person support; (S3) Learning collaborative, (S2) in-person support; Experimental: (S1) E-support, (S2) in-person support, (S3) Learning collaborative
Behavioral: Learning collaborative — Access to an online information-sharing portal, monthly newsletter, annual face-to-face half day conference
  Arms: (S1) E-support, (S3) Learning collaborative; (S3) Learning collaborative; (S3) Learning collaborative, (S2) in-person support; Experimental: (S1) E-support, (S2) in-person support, (S3) Learning collaborative

SUMMARY:
This project compares four SAGE implementation strategies to evaluate effectiveness in implementation, sustainability, cost, and child health outcomes. Using the CFIR and MOST frameworks, the investigators will analyze key components to identify the most efficient and scalable strategies. Data will come from ECE site audits, surveys, social network analysis, and child health assessments. Findings will inform sustainable, cost-effective approaches to improve early childhood nutrition and physical activity.

DETAILED DESCRIPTION:
The overall objective of this project is to compare how four different SAGE implementation strategies impact measures of implementation (primary), sustainability (secondary), cost and child health outcomes (secondary). Strategies the investigators will compare include (1) SAGE (garden + online curriculum + materials box) vs. SAGE plus e-support implementation package (text messages + newsletters + hotline), (2) SAGE with no in person support and training vs. SAGE with in person support and training, and (3) SAGE usual activities vs. SAGE with a ECE virtual learning collaborative to share SAGE implementation experiences and strategies with other ECE sites and community partners. The investigators will (Aim 1) apply the Consolidated Framework for Implementation Research (CFIR) to identify inner and outer setting characteristics that hinder or facilitate SAGE implementation to tailor support strategies for local context; (Aim 2) use the Multiphase Optimization Strategy (MOST) framework to analyze SAGE implementation strategy components to determine the most efficient and effective combination of strategies across contexts; and (Aim 3) investigate the potential for sustainability, costs and cost effectiveness outcomes that may influence implementation strategies and their effect on locomotor skills and nutrition effectiveness outcomes. In Aim 1 (MOST screening), the investigators will measure ECE site and teacher characteristics via an in person visual assessment and a teacher and director survey (inner setting). The investigators will also complete a social network analysis of ECE personnel. With this information the investigators will use an implementation mapping process to collaboratively develop and finalize implementation strategies. In Aim 2 (MOST refine), 32 existing SAGE ECE sites will be pair matched by degree of individual implementation and site characteristics (size, enrollment) assessed in aim 1, and assigned to one of eight implementation strategy combinations to a full factorial model. Sites will be assessed at the beginning and ending of the academic year with site audits, parent and teacher surveys, and non-invasive child fitness, physical activity, veggiemeter and eating in the absence of hunger measures. For Aim 3, (MOST refine) the potential for sustainability, costs and cost effectiveness ratio for each of the strategies will be calculated from a payer and societal perspective to determine which implementation strategy or combination of strategies may be most scalable.

ELIGIBILITY:
Inclusionary criteria:

ECE personnel, child, or parent of enrolled eligible ECE site Provided consent and/or assent

Exclusion criteria:

Allergy or condition which prohibits participation in garden-based curricula

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 871 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Implementation | Baseline, 6 mos post-test, 16 months follow up
  Proportion of teachers who rate SAGE as acceptable, appropriate, and feasible to implement.
  Proportion of teachers completing at least 70% of curriculum activities as measured by weekly fidelity checklists.

SECONDARY OUTCOMES:
Locomotor skills | Baseline, 6 mos post-test, 16 months follow up
  The Children's Activity and Movement in Preschool Study Motor Skills Protocol (CMSP) measures six developmentally appropriate skills (run, broad jump, slide, gallop, leap, and hop). The locomotor subscale ranges from 0 to 64 skill components, with a higher score indicating better locomotor skills.
Veggiemeter | Baseline, 6 mos post-test, 16 months follow up
  An objective assessment of fruit and vegetable intake through a direct measure of dietary carotenoids
Eating in the absence of hunger | Baseline, 6 mos post-test, 16 mos follow up
  Children are tested on consumption of sweet and salty snacks immediately following a meal to determine whether they eat in the absence of hunger
Moderate to vigorous physical activity | Baseline, 6 mos post-test, 16 mos follow up
  Children wear a small accelerometer device to measure MVPA for a six hour period on consecutive days during the ECE day

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected as part of this project will be de-identified and made available on public websites that may be shared with investigators working under an institution with a Federal Wide Assurance (FWA). As there is no specific data sharing repository for the funding agency, the investigators will identify possible other repositories that may be appropriate to use. For whatever NIH-funded repository is advised to be used, the investigators acknowledge that this repository will have policies and procedures in place that will provide data access to qualified researchers, consistent with NIH data sharing policies and applicable laws and regulations. Data will be deposited to the repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and statistical Analysis Plan will be available by January 2028 with no end date.
Access Criteria: Data could be used for secondary study purposes such as finding additional relationships related to implementation and sustainability of garden based education in early care and education. Data will be openly available.